CLINICAL TRIAL: NCT00710775
Title: Temporary Intra-operative Placement of HLT Percutaneous Aortic Valve
Brief Title: Heart Leaflet Technologies Valve Study
Acronym: HLT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Cardiologico Monzino (Other)
Responsible Party: Paolo Biglioli, Prof., Centro Cardiologico Monzino-University of Milan
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: R78- CCM S80/507
Record Dates: First submitted 2008-06-27; First posted 2008-07-04 (Estimated); Last update posted 2009-10-12 (Estimated); Status verified 2008-05

CONDITIONS: Aortic Valve Stenosis; Endovascular Aortic Valve Replacement
Keywords: Aortic valve stenosis; Heart surgery; Endovascular techniques
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Patients undergoing surgical aortic valve replacement on cardiopulmonary bypass.
  Interventions: Procedure: surgical replacement of the aortic stenotic valve

INTERVENTIONS:
Procedure: surgical replacement of the aortic stenotic valve — Prior to surgical removal of the aortic valve, the native valve will be dilated under direct vision of the surgeon using a standard valve dilation balloon. The HLT valve will be loaded into a short version of the delivery catheter system and the catheter will be passed across the native valve.Measurements will be taken of the device relative to the anatomic structures of the heart. Once complete, the implant is removed from the native valve and the surgical valve replacement procedure is completed.
  Other Names: AVR (aortic valve replacement)

SUMMARY:
The study will be conducted in patients who are undergoing surgical aortic valve replacement on cardiopulmonary bypass. Following surgical access of the native aortic valve and prior to removal of the valve, the native valve will be dilated using a standard valve dilation balloon. The Heart Leaflet Technologies(HLT- Heart Leaflet Technologies Inc.) aortic valve device will be released in the native valve and measurements will be taken of the device relative to the anatomic structures of the heart. Once completed, the implant is removed from the native valve and the surgical valve replacement procedure is completed.

The purpose of this study is to confirm that the dimensions of the HLT valve are appropriate for patients with aortic valve stenosis.

DETAILED DESCRIPTION:
Aortic valve stenosis is a disease in which the leaflets of the aortic valve become scarred and calcified. This leads to a severe narrowing of the valve orifice, which causes chest pain, heart failure and eventually death. The condition is currently treated with open chest surgical valve replacement on cardiopulmonary bypass. Heart Leaflet Technologies has developed an aortic valve prosthesis that can be delivered to the stenotic aortic valve through a catheter inserted in the femoral artery.

The purpose of this study is to confirm that the dimensions of the HLT valve are appropriate for patients with aortic valve stenosis. There is no animal model of aortic valve stenosis. Heart Leaflet Technologies has performed extensive device geometry and deployment testing on fixed cadaveric hearts with calcified cusps and aortic stenosis. HLT has also performed a number of preclinical animal experiments to verify deliverability and device function in vivo.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing aortic valve replacement for aortic valve stenosis with a preoperative valve area < 0.9 cm2.
2. A preoperative echocardiogram where the aortic annulus diameter can be measured and is between 19 and 25 mm internal diameter.
3. Age 75 to 80 years

Exclusion Criteria:

1. Emergency valve surgery
2. Significant ascending aortic disease (atheroma, extensive calcification, dissection) as assessed by the operating surgeon
3. Ostial coronary obstruction > 25% diameter stenosis

Ages: 75 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2007-11; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
geometrical evaluation of HLT pliability to patient's native aortic valve | during surgery procedure

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Biglioli, MD, Principal Investigator — Centro Cardiologico Monzino-University of Milan
Locations (1):
- Centro Cardiologico Monzino- University of Milan, Italy, Milan, Italy

REFERENCES:
- [Background] Ghanbari H, Kidane AG, Burriesci G, Bonhoeffer P, Seifalian AM. Percutaneous heart valve replacement: an update. Trends Cardiovasc Med. 2008 May;18(4):117-25. doi: 10.1016/j.tcm.2008.02.002. PMID 18555184
- [Background] Webb JG. Percutaneous aortic valve replacement. Curr Cardiol Rep. 2008 Mar;10(2):104-9. doi: 10.1007/s11886-008-0019-z. PMID 18417010
- [Background] Rosengart TK, Feldman T, Borger MA, Vassiliades TA Jr, Gillinov AM, Hoercher KJ, Vahanian A, Bonow RO, O'Neill W; American Heart Association Council on Cardiovascular Surgery and Anesthesia; American Heart Association Council on Clinical Cardiology; Functional Genomics and Translational Biology Interdisciplinary Working Group; Quality of Care and Outcomes Research Interdisciplinary Working Group. Percutaneous and minimally invasive valve procedures: a scientific statement from the American Heart Association Council on Cardiovascular Surgery and Anesthesia, Council on Clinical Cardiology, Functional Genomics and Translational Biology Interdisciplinary Working Group, and Quality of Care and Outcomes Research Interdisciplinary Working Group. Circulation. 2008 Apr 1;117(13):1750-67. doi: 10.1161/CIRCULATIONAHA.107.188525. Epub 2008 Mar 10. PMID 18332270